CLINICAL TRIAL: NCT04926077
Title: Validation of the DreamKit Plethysmography-derived Respiratory Effort Signal Against Esophageal Pressure
Brief Title: DreamKit Respiratory Effort Signal Validation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Clinical & Medical Affairs Global (Industry)
Collaborators: Pulmonary Critical Care Associates of Baltimore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SRC_SLE_SparkleEP2_2021_11315
Record Dates: First submitted 2021-06-08; First posted 2021-06-14 (Actual); Results first posted 2022-11-30 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Sleep Apnea, Obstructive; Sleep Apnea, Central
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea, Central

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Validation Arm (Experimental): Participants will wear the DreamKit device (test device) while instrumented with an esophageal manometry catheter (reference standard) to record respiratory effort.
  Interventions: Device: DreamKit

INTERVENTIONS:
Device: DreamKit — The DreamKit device is a single-use device intended to aid the diagnosis of sleep-disordered breathing; however, this study is intended only to validate the respiratory effort signal and does not assess diagnostic performance.

SUMMARY:
This study has been developed in order to demonstrate the validity of the DreamKit respiratory effort signal.

DETAILED DESCRIPTION:
The rationale for undertaking this study is to demonstrate the agreement between the respiratory effort signal amplitude derived from DreamKit vs. the gold-standard esophageal manometry. Data collection will be completed within a single visit, in which participants will undergo simultaneous measurement using the DreamKit device and esophageal manometry. Data collection will be completed during wakefulness, while participants undergo a series of breathing maneuvers.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years;
* Fluent in English;
* Able to provide informed consent.

Exclusion Criteria:

* Contraindication to esophageal pressure monitoring, including a sensitive gag reflex (determined by a positive response to the screening question "do you sometimes or often gag while brushing your teeth?"), dysphagia, nasal obstruction, and/or esophageal disorder likely to impact placement of the balloon;
* Pregnancy or planned pregnancy during the study (self-reported);
* History of allergic reactions to medical adhesives;
* Known allergy to lidocaine;
* Known seizure disorder;
* Severe medical condition (controlled or uncontrolled) impacting breathing including neuromuscular disease, chronic obstructive pulmonary disease, respiratory failure or insufficiency, or requirement for oxygen therapy;
* Chronic cardiopulmonary or renal disease, including a history of irregular heart rhythms or dyspnea;
* At risk for excessive bleeding including use of anticoagulants;
* An employee, or spouse of an employee, of a company that designs, sells, or manufactures sleep related products (including Philips);
* An employee, or spouse of an employee, of Pulmonary & Critical Care Associates of Baltimore.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-06-22 (Actual); Primary Completion 2021-10-07 (Actual); Study Completion 2021-10-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Schwartz, MD, Principal Investigator — Pulmonary Critical Care Associates of Baltimore
Locations (1):
- Pulmonary and Critical Care Associates of Baltimore, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Validation Arm
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All participants that signed a consent form.
Arm/Group | Validation Arm
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.3 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 11
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 27.2 (6.7)

OUTCOME MEASURES:

1. Primary Outcome: Breath Amplitude Correlation
Description: The primary endpoint is the intraclass correlation coefficient (ICC) of the peak-to-peak breath amplitude sequences extracted from the DreamKit and esophageal manometry respiratory effort signals during periods of occluded inspiration, end-expiratory breath holds, increased inspiratory resistance, increased expiratory resistance, and unresisted shallow breathing. The DreamKit Home Sleep Test device's effort signal is an uncalibrated signal. The amplitudes derived from the DreamKit Home Sleep Test device's effort signal were scaled for each subject to have the same variance across all tested breathing maneuvers. The lower-bound of the CI was compared against a target of 0.5.
Time Frame: Baseline
Population: 1 participant was excluded from the data analysis due to bad signal quality indicated by the DreamKit Home Sleep Test device.
Measure: Number (95% Confidence Interval); unit: ICC the aggregated signal amplitudes
Arm/Group | Validation Arm
Number analyzed (Participants) | 10
ICC the aggregated signal amplitudes | .66 [.64 to .67]

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Validation Arm
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-24): https://cdn.clinicaltrials.gov/large-docs/77/NCT04926077/Prot_SAP_000.pdf